CLINICAL TRIAL: NCT03614312
Title: Epigenetic Mechanisms Underlying Trophoblast Syncytialization
Brief Title: Placenta Development Study
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 206617
Record Dates: First submitted 2018-03-05; First posted 2018-08-03 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Placenta, umbilical cord, and cord blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BMI 18-25 Pregnant Women: BMI 18-25 less than 36 weeks pregnant

SUMMARY:
This study will help us learn more about how the placenta develops.

DETAILED DESCRIPTION:
The primary purpose of this study is to understand the epigenetic signaling events in placental trophoblast development.

ELIGIBILITY:
Inclusion Criteria:

* BMI - 18-25 kg/m2
* at least 18 years of age
* singleton pregnancy
* less than 36 weeks and plan to deliver in the Little Rock/North Little Rock Area

Exclusion Criteria:

* Women with pre-existing medical conditions (e.g. diabetes, hypertension, pre-eclampsia, STD, gestational diabetes)
* Women who are using recreational drugs, tobacco, or alcohol during their pregnancy.
* Women who plan on keeping their placenta following delivery for non-medical reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Number of participants that placental syncytial fusion involves epigenetic changes in histone modifications | 40 weeks
  Number of participants that histone acetyltransferases eszymes, CBP and p300 affect syncytial fusion

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No